CLINICAL TRIAL: NCT01730768
Title: A 12 Week, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Effects of Once Daily Doses of AQW051 on Cognition, in Stable Schizophrenia Patients
Brief Title: A Study to Evaluate the Effects of Once Daily Doses of AQW051 on Cognition, in Stable Schizophrenia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A2207
Record Dates: First submitted 2012-09-06; First posted 2012-11-21 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia, chronic stable schizophrenia, cognition, memory, visual learning, CogState
MeSH Terms: conditions — Schizophrenia; Spatial Learning | interventions — 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AQW051 10 mg/day (Experimental): Two 5mg AQW051 capsules will be taken orally daily by patients from Day 1 until Day 84.
  Interventions: Drug: AQW051
- Placebo to AQW051 (Placebo Comparator): Matching placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQW051
  Arms: AQW051 10 mg/day
Drug: Placebo
  Arms: Placebo to AQW051

SUMMARY:
This is a study in chronic stable Schizophrenia with the purpose to answer the question of whether agonism of the nicotinic alpha7 receptor is capable of enhancing cognition in a well defined chronic stable patient population treated with antipsychotics as standard of care, and thus to support the future development of AQW051 for the treatment of cognitive impairment associated with Schizophrenia (CIAS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Symptomatically stable and currently treated with a stable regimen for at least 3 (three) months prior to dosing with one of the following second generation of antipsychotics: risperidone, paliperidone, quetiapine, ziprasidone, aripiprazole.
* Specific cognitive impairment
* Smokers and non-smokers

Exclusion Criteria:

* Current treatment with an anticholinergic or other agent known to adversely interfere with the cholinergic system, and/ or treatment with cholinesterase inhibitor within the last three (3) months prior to dosing.
* Current treatment with conventional antipsychotics (e.g fluphenazine, haloperidol) or clozapine.
* History of neuroleptic malignant syndrome.
* Diagnosis of substance abuse (other than nicotine) within the last month and alcohol or substance dependence (other than nicotine) within the last 6 months.
* Score 4 or 5 on the Suicidal Ideation item or any "yes" on the Suicidal Behavior item of the CSSR-S that is related to suicidal behavior occurring during the last 2 years

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual learning and memory at 4 weeks | 4 weeks
  The primary objective is to evaluate the pro-cognitive effects of AQW051 in a chronic stable schizophrenic patient population at week 4 as measured by the absolute change from baseline in CPAL number of errors (CogState battery) at week 4.

SECONDARY OUTCOMES:
Effect on cognitive function after 12 weeks of treatment - CogState test battery. | Baseline, 12 weeks
  Change from baseline will be analyzed using a mixed model for repeated measures, including baseline value as covariate, time (timepoint), treatment as fixed effects and treatment*time interaction term and patient as random effect. Appropriate contrasts will be used to compare treatments at each timepoint.
Effect on cognitive function after 12 weeks of treatment - MCCB | Baseline, 12 weeks
  Change from baseline will be analyzed using a mixed model for repeated measures, including baseline value as covariate, time (timepoint), treatment as fixed effects and treatment*time interaction term and patient as random effect. Appropriate contrasts will be used to compare treatments at each timepoint.
Number of patients with adverse events | 12 weeks
  Summarized statistics on adverse events will be reported under categories such as total adverse events, serious adverse events and death.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Novartis Investigative Site, Garden Grove, California
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, National City, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Pico Rivera, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Miramar, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marlton, New Jersey
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Irving, Texas

REFERENCES:
- See also: Results for CAQW051A2207 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12903